CLINICAL TRIAL: NCT03627624
Title: Minimal Clinically Important Difference in 30 Second Sit-to-stand Test After Pulmonary Rehabilitation in Patients With COPD
Brief Title: MCID in 30 STS Test After PR in COPD Patients
Acronym: COPD
Status: Completed | Type: Observational
Sponsor: elisabetta zampogna (Other)
Collaborators: University of Parma (Other); Ospedale Civico, Lugano (Other Government); Università degli Studi dell'Insubria (Other)
Responsible Party: Sponsor-Investigator, elisabetta zampogna, sub-investigator, Maugeri Foundation
Organization: Maugeri Foundation (Other)
Other Study IDs: Maugeri2
Record Dates: First submitted 2018-07-06; First posted 2018-08-13 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: COPD
Keywords: MCID; 30 STS test; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonary rehabilitation — Stable COPD inpatients undergoing 30-STST and 6-minute walk test (6MWT) before and after PR were included. Responsiveness to PR was determined by pre-to-post PR (Δ) evaluation of 30-STST.

SUMMARY:
The sit-to-stand test (STST) is a feasible alternative for measuring peripheral muscle strength of the lower limbs.

Our aim was to evaluate, in Chronic Obstructive Pulmonary Disease (COPD) patients, the minimal clinically important difference (MCID) of 30-second STST (30-STST) after pulmonary rehabilitation (PR).

Stable COPD inpatients undergoing 30-STST and 6-minute walk test (6MWT) before and after PR were included. Responsiveness to PR was determined by pre-to-post PR (Δ) evaluation of 30-STST. The MCID was evaluated using an anchor-based method.

DETAILED DESCRIPTION:
The sit-to-stand test (STST) is a feasible alternative for measuring peripheral muscle strength of the lower limbs used as standard test at the beginning and at the end of pulmonary rehabilitation programme.

Our aim was to retrospectively evaluate, in Chronic Obstructive Pulmonary Disease (COPD) patients, the minimal clinically important difference (MCID) of 30-second STST (30-STST) after pulmonary rehabilitation (PR).

Stable COPD inpatients undergoing 30-STST and 6-minute walk test (6MWT) before and after PR were included. Responsiveness to PR was determined by pre-to-post PR (Δ) evaluation of 30-STST. The MCID was evaluated using an anchor-based method.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis for COPD according to the GOLD criteria.
* no exacerbations over the previous four weeks

  - Page 3 of 3 -
* completing PR program
* smoking history ≥10 pack years
* regular treatment with inhaled bronchodilators and inhaled steroids

Exclusion Criteria:

* any unstable medical condition
* Contraindications for participation in the PR program included musculoskeletal disorders, malignant diseases, unstable cardiac condition, and lack of adherence to the program -

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We examined 96 patients with COPD who attended an inpatient PR program. All patients had a diagnosis for COPD according to the GOLD criteria.Patients who had acute exacerbation over the previous four weeks were excluded. Patients who did not complete the PR program, for intercurrent COPD exacerbation, or any unstable medical condition, were also excluded. Contraindications for participation in the PR program included musculoskeletal disorders, malignant diseases, unstable cardiac condition, and lack of adherence to the program. All patients had smoking history ≥10 pack years and received regular treatment with inhaled bronchodilators and inhaled steroids according to current guidelines for their disease stage.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
30 STS test | 21 days
  Minimally clinically important difference

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof, Study Chair — Maugeri Foundation
Locations (2):
- ICS Maugeri, Tradate, Varese, Italy
- EOC, Novaggio, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Debigare R, Cote CH, Maltais F. Peripheral muscle wasting in chronic obstructive pulmonary disease. Clinical relevance and mechanisms. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1712-7. doi: 10.1164/ajrccm.164.9.2104035. No abstract available. PMID 11719314
- [Background] Skeletal muscle dysfunction in chronic obstructive pulmonary disease. A statement of the American Thoracic Society and European Respiratory Society. Am J Respir Crit Care Med. 1999 Apr;159(4 Pt 2):S1-40. doi: 10.1164/ajrccm.159.supplement_1.99titlepage. No abstract available. PMID 10194189
- [Background] Spruit MA, Gosselink R, Troosters T, De Paepe K, Decramer M. Resistance versus endurance training in patients with COPD and peripheral muscle weakness. Eur Respir J. 2002 Jun;19(6):1072-8. doi: 10.1183/09031936.02.00287102. PMID 12108859
- [Background] Ortega F, Toral J, Cejudo P, Villagomez R, Sanchez H, Castillo J, Montemayor T. Comparison of effects of strength and endurance training in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2002 Sep 1;166(5):669-74. doi: 10.1164/rccm.2107081. PMID 12204863
- [Background] Troosters T, Probst VS, Crul T, Pitta F, Gayan-Ramirez G, Decramer M, Gosselink R. Resistance training prevents deterioration in quadriceps muscle function during acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 May 15;181(10):1072-7. doi: 10.1164/rccm.200908-1203OC. Epub 2010 Feb 4. PMID 20133927
- [Background] Simpson K, Killian K, McCartney N, Stubbing DG, Jones NL. Randomised controlled trial of weightlifting exercise in patients with chronic airflow limitation. Thorax. 1992 Feb;47(2):70-5. doi: 10.1136/thx.47.2.70. PMID 1549826
- [Derived] Zanini A, Crisafulli E, D'Andria M, Gregorini C, Cherubino F, Zampogna E, Azzola A, Spanevello A, Schiavone N, Chetta A. Minimum Clinically Important Difference in 30-s Sit-to-Stand Test After Pulmonary Rehabilitation in Subjects With COPD. Respir Care. 2019 Oct;64(10):1261-1269. doi: 10.4187/respcare.06694. Epub 2019 Jul 3. PMID 31270178